CLINICAL TRIAL: NCT06413017
Title: Nimotuzumab Combined With Immune Checkpoint Inhibitors for the Treatment of Advanced Liver Cancer After First Line Treatment Failure ，a Prospective， Open Label，Single Arm，Phase II Trail
Brief Title: Nimotuzumab Combined With ICIs for the Treatment of Advanced Liver Cancer After First Line Treatment Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Jihui Hao, Chief physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nim-PC-7
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: HCC
MeSH Terms: interventions — nimotuzumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimtuzumab combined ICIs (Experimental): Patients will be treated with nimotuzumab combined immune checkpoint inhibitors treatment
  Interventions: Drug: Nimotuzumab; Drug: ICIs(Immune checkpoint inhibitors)

INTERVENTIONS:
Drug: Nimotuzumab — Nimtuzumab：400mg,i.v.,once a week,until tumor progression、Death or untalerable toxicity
  Other Names: h-R3
Drug: ICIs(Immune checkpoint inhibitors) — Use it as it is describe in the instructions from the specification
  Other Names: PD-1 or PD-L1

SUMMARY:
This is a phase II, open-label, single-arm clinical study of nimotuzumab in combination with immune checkpoint inhibitors in patients with advanced liver cancer who have failed first-line therapy

DETAILED DESCRIPTION:
This study is a prospective, single-arm study, and plans to include 30 patients with hepatocellular carcinoma who do not respond to first-line therapy with a protoPD-1 (or PD-L1) inhibitor in combination with nimotuzumab in the posterior line, and receive nimotuzumab 400mg, D1, QW in combination with PD-1 (or PD-L1) inhibitor in the later line of treatment until disease progression and intolerable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed advanced hepatocellular carcinoma (HCC), or The clinical diagnosis meets the American Association of Liver Diseases (AASLD) diagnostic criteria for hepatocellular carcinoma；
* Prior experience of targeted, immune, progression after conventional therapy, or intolerance (including TKIs,ICIs, chemotherapy, VEGF monoclonal antibody, or ICIs in combination with TKIs/VEGFs monoclonal antibody/chemotherapy)；
* Child-Pugh liver function rating within 7 days prior to the first dose of study drug: Grade A or better grade B (≤ 7 points) ;
* Phase B or C as assessed by BCLC; or Phase III as assessed by CNLC;
* Within 4 weeks prior to the first dose, at least one measurable target lesion remained according to mRECIST v1.1；
* EGFR postive and RAS wildtype；

Exclusion Criteria:

* Dignosised as hepatic cholangiocarcinoma, mixed cell carcinoma, or fibrolamellar cell carcinoma；
* History of hepatic encephalopathy within 6 months prior to the first dose of this study；
* Portal hypertension with endoscopic red signs, or those who are considered by the investigator to be at high risk of bleeding or who have had esophageal or gastric variceal bleeding within 6 months prior to the first dose；
* Symptomatic brain or meningeal metastases (unless patient is treated> 3 months, no evidence of progression on imaging within 4 weeks prior to treatment, and tumor-related clinical symptoms is stable)

Ages: 17 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR（Objtective reseponse rate） | up to 24 month
  （Objtective reseponse rate）

SECONDARY OUTCOMES:
OS（overall survival） | up to 24 month
  Time from the first dose to death
PFS（pregression free survival） | up to 24 month
  time form fist dose to tumor progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Dr, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No